CLINICAL TRIAL: NCT06942273
Title: Analysis of Hyperthermia as a Complementary Treatment to Evidence-based Clinical Intervention in Subjects With Carpal Tunnel Syndrome: a Double-blind Randomized Clinical Trial.
Brief Title: Analysis of Hyperthermia as a Complementary Treatment to Evidence-based Clinical Intervention in Subjects With Carpal Tunnel Syndrome:
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 45/2025
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Carpal Tunnel Syndrome (CTS); Hyperthermia; Frequency of Therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Hyperthermia | interventions — Diathermy; Exercise; Splints

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hyperthermia 2 times per week (Experimental)
  Interventions: Radiation: hyperthermia; Other: physical exercise; Other: splint
- Hyperthermia 3 times per week (Experimental)
  Interventions: Radiation: hyperthermia; Other: physical exercise; Other: splint
- Non-hyperthermia 2 times per week (Experimental)
  Interventions: Other: physical exercise; Other: splint
- Non-hyperthermia 3 times per week (Experimental)
  Interventions: Other: physical exercise; Other: splint

INTERVENTIONS:
Radiation: hyperthermia — hyperthermia over the carpal tunnel area and adjacent areas
  Arms: Hyperthermia 2 times per week; Hyperthermia 3 times per week
Other: physical exercise — Performing therapeutic physical exercise focused on the flexor muscles of the hand and neural stretching
Other: splint — imposition of a night splint

SUMMARY:
This project aims to analyze the use of hyperthermia within a treatment protocol for Carpal Tunnel Syndrome (CTS), as well as to determine the difference between two and three sessions per week. Study participants will be divided into four intervention groups: the first will receive two sessions per week for a period of six months, while the second will receive three sessions per week for the same period. The treatment protocol will consist of therapeutic physical exercise focused on the hand flexor muscles and neural stretching, the application of hyperthermia to the carpal tunnel and adjacent areas, and the use of a night splint. The third and fourth intervention groups will receive the same treatment as mentioned above, but without hyperthermia. The third group will receive three sessions per week, while the second group will receive two sessions per week. Two different types of measurement variables will be used: objective variables will be used to measure hand flexor muscle strength and wrist free range of motion. Subjective variables will also be used through validated questionnaires covering physical activity, perceived functional limitations, upper limb functional assessment, neuropathic pain, and a visual analogue scale for pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis confirmed by performing an electromyography of Carpal Tunnel Syndrome
* Have not yet received physiotherapy treatment.

Exclusion Criteria:

* Have undergone surgery.
* Those who refuse to participate in this study.
* Patients with muscle atrophy due to CTS.
* Medical conditions that are contraindications for hyperthermia therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) | Baseline and up to one year
  Minimum: 19. Maximum: 95. A higher score indicates a higher degree of disability
Disabilities of arm, shoulder and hand (DASH) | Baseline and up to one year
  Minimum: 30 points. Maximum: 150 points A higher score indicates a higher intensity of symptoms
Neuropathic Pain Scale (DN4) | Baseline and up to one year
  Minimum: 0 Maximum: 10 The diagnosis of neuropathic pain is established with a total scale of 4 out of 10
International Physical Activity Questionnaire (IPAQ) | Baseline and up to one year
  9 items. Minimum: 9 Maximum: 36 A higher score indicates a sedentary life
Visual Analogue Scale (VAS) | Baseline and up to one year
  Minimum: 1 Maximum: 10 A higher score indicates a higher intensity of pain
Hand grip strength | Baseline and up to one year
  A handheld dynamometer will be used and three consecutive measurements will be obtained with the patient sitting and the elbow flexed at 90 degrees and in a neutral position.
WRIST JOINT RANGE OF MOBILITY | Baseline and up to one year
  With the patient seated in a relaxed position, the various free movements of the wrist joint will be assessed bilaterally using an electronic goniometer. To do this, the goniometer will be placed on the dorsal side of the wrist, with the proximal part on the midline between the radius and ulna and the distal part on the third metacarpal. Flexion, extension, and radial and ulnar deviation ranges will be assessed, both with the elbow flexed and extended.
WRIST FLEXION EVALUATION TEST | Baseline and up to one year
  With the patient seated in a relaxed position, wrist flexion will be tested in isometric contraction, both with the hand open and closed, and with the wrist in a neutral position. The therapist will manually resist wrist flexion from the hand area. This test will be performed three times in a row with the hand open, followed by a five-minute rest and then repeating the procedure, this time with the hand open. This measurement will be taken with the elbow flexed or extended.